CLINICAL TRIAL: NCT03739528
Title: An International, Multicenter, Randomized, Blinded-assessor, Parallel-group Clinical Study Comparing Eye Drops of Combined LEvofloxAcin + DExamethasone foR 7 Days Followed by Dexamethasone Alone for an Additional 7 Days vs. Tobramycin + Dexamethasone for 14 Days for the Prevention and Treatment of Inflammation and Prevention of Infection Associated With Cataract Surgery in Adults - LEADER 7
Brief Title: Levo-Dexa vs. Tobra+Dexa for Prevention and Treatment of Inflammation and Prevention of Infection in Cataract Surgery
Acronym: LEADER7
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NTC srl (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LEVODESA_04-2017
Record Dates: First submitted 2018-11-09; First posted 2018-11-14 (Actual); Results first posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Levofloxacin; Tobramycin, Dexamethasone Drug Combination

STUDY DESIGN:
Intervention Model Description: A randomized, parallel-group study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levofloxacin + Dexamethasone followed by dexamethasone (Experimental): Levofloxacin 5 mg/ml+Dexamethasone 1 mg/ml (7 days,1 drop/4 times a day) followed by dexamethasone 1 mg/ml (7 days,1 drop/4 times a day).
  Interventions: Drug: Levofloxacin + dexamethasone followed by dexamethasone
- Tobramycin + dexamethasone (Active Comparator): Tobramycin + dexamethasone (14 days, 1 drop/4 times a day).
  Interventions: Drug: Tobramycin + Dexamethasone

INTERVENTIONS:
Drug: Levofloxacin + dexamethasone followed by dexamethasone — Levofloxacin + dexamethasone ophthalmic solution for 7 days, 1 drop - 4 times a day, followed by dexamethasone ophthalmic suspension (Maxidex®) for an additional 7 days, 1 drop - 4 times a day.
  Other Names: Levofloxacin + dexamethasone followed by Maxidex
  Arms: Levofloxacin + Dexamethasone followed by dexamethasone
Drug: Tobramycin + Dexamethasone — Tobramycin + dexamethasone ophthalmic suspension (Tobradex®) for 14 days, 1 drop - 4 times a day.
  Other Names: Tobradex
  Arms: Tobramycin + dexamethasone

SUMMARY:
The purpose of this study is to demonstrate the non-inferiority of the study treatment (combined levofloxacin + dexamethasone eye drops) followed by dexamethasone eye drops alone vs. standard treatment in the prevention and treatment of postoperative ocular inflammation and prevention of infection.

DETAILED DESCRIPTION:
In clinical practice, topical treatment following cataract surgery is frequently administered using a combination between an antibiotic and a corticosteroid to promote patient adherence to therapy and to obtain both prevention of infection and treatment of post-surgical inflammation.

The combination of tobramycin and dexamethasone is among the most widely used combinations, however, treatment duration and the need for tapering posology over several weeks may favour the development of bacterial resistance. The study treatment associating a broad-spectrum antibiotic with a highly effective corticosteroid that can be used for a short period of time (one week) is therefore of considerable interest.

The aim of this study is to evaluate the non-inferiority of the study treatment, used for a limited period of time and followed by dexamethasone alone, compared to standard treatment in preventing and treating ocular inflammation and in preventing post-operative infection while limiting the emergence of antibiotic resistance.

ELIGIBILITY:
Inclusion Criteria prior to surgery:

1. Signed written informed consent
2. Male or female, age ≥40 years
3. Scheduled senile or presenile cataract surgery
4. Willing to interrupt the use of contact lenses for the entire duration of the study
5. Able and willing to follow study procedures
6. Female patients must be postmenopausal, surgically sterile or must agree to use an effective method of contraception

   Inclusion criteria following surgery:
7. Surgery completed without complications

Exclusion Criteria:

1. Ocular conditions that at the discretion of the Investigator may interfere with the efficacy and/or safety evaluations
2. Patients undergoing bilateral cataract surgery
3. Patients under treatment with prostaglandin analogues or intravitreal injections of anti-vascular endothelial growth factor (VEGF) drugs
4. Systemic diseases that may interfere with the results of the study
5. Any condition that could interfere with correct instillation of eye drops
6. Ocular surgery in the study eye (including laser surgery) in the 3 months before screening
7. Monocular patients
8. Visual Acuity < 20/80 of the contralateral eye measured as ETDRS or Snellen
9. Contraindications to ocular treatment with Tobradex®, Maxidex® or levofloxacin/dexamethasone
10. Hypersensitivity to the study product or its excipients
11. Participation in other clinical studies within at least 5 half-lives of the Investigational Medicinal Product (IMP) used in the previous studies
12. Pregnancy or breastfeeding

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 808 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Bandello, Prof., Principal Investigator — Ospedale San Raffaele IRCCS S.r.l.
Locations (57):
- Italy (57):
  - A.O.U. Osp. Riuniti Umberto I - G.M. Lancisi - G. Salesi - Università degli Studi di Ancona, Ancona, AN
  - Ospedale della Murgia "Fabio Perinei" di Altamura, Altamura, BA
  - A.O.U. Policlinico Consorziale di Bari, Bari, BA
  - ASL Bari - Ospedale "Di Venere" - Carbonara di Bari, Bari, BA
  - Cliniche Gavazzeni S.p.A. - Humanitas Gavazzeni di Bergamo, Bergamo, BG
  - A.O.U. di Bologna - Policlinico S. Orsola-Malpighi di Bologna, Bologna, BO
  - Policlinico S. Orsola-Malpighi di Bologna, Bologna, BO
  - ASST degli Spedali Civili di Brescia - P.O. Spedali Civili di Brescia, Brescia, BS
  - ASST Franciacorta - P.O. di Chiari, Chiari, BS
  - P.O. Ospedale Clinicizzato SS. Annunziata di Chieti, Chieti, CH
  - Ospedale Valduce di Como, Como, CO
  - A.O.U. Policlinico Vittorio Emanuele - P.O. Gaspare Rodolico - Università degli Studi di Catania, Catania, CT
  - Policlinico G.B. Morgagni di Catania - Casa di Cura s.r.l., Catania, CT
  - A.O. Mater Domini di Catanzaro - Università degli Studi Magna Graecia di Catanzaro, Catanzaro, CZ
  - IRCCS Casa Sollievo della Sofferenza di San Giovanni Rotondo, San Giovanni Rotondo, FG
  - A.O.U. Careggi di Firenze, Florence, FI
  - IRCCS Ospedale Policlinico San Martino di Genova, Genova, GE
  - Ospedale Policlinico San Martino - Università degli Studi di Genova, Genova, GE
  - Fatebenefratelli - Ospedale "Sacra Famiglia" di Erba, Erba, LC
  - Az. USL Toscana Nord Ovest - Ospedale della Versilia, Lido di Camaiore, LU
  - AUSL Toscana Nord Ovest - P.O. San Luca di Lucca, San Filippo, LU
  - A.O.U. Policlinico "G. Martino" di Messina, Messina, ME
  - ASP di Messina - P.O. "Giuseppe Fogliani" di Milazzo, Milazzo, ME
  - ASST Ovest Milanese - Ospedale Civile di Legnano, Legnano, MI
  - IRCCS Ca' Granda Ospedale Maggiore Policlinico di Milano, Milan, MI
  - Gruppo Multimedica - Ospedale San Giuseppe di Milano, Milan, MI
  - Ospedale San Raffaele IRCCS S.r.l., Milan, MI
  - ASST Fatebenefratelli Sacco - Università degli Studi di Milano - Ospedale L. Sacco, Milan, MI
  - IRCCS Istituto Clinico Humanitas di Rozzano, Rozzano, MI
  - ASST di Melegnano e della Martesana - Ospedale di Vizzolo Predabissi, Vizzolo Predabissi, MI
  - A.O.U. Policlinico di Modena - Università degli Studi di Modena e Reggio Emilia, Modena, MO
  - Ospedale di Sassuolo, Sassuolo, MO
  - Centro Polispecialistico Monterosso di Carrara, Carrara, MS
  - A.O.U. Policlinico "P. Giaccone" di Palermo, Palermo, PA
  - A.O. "Ospedali Riuniti Villa Sofia-Cervello" di Palermo - P.O. "Villa Sofia" di Palermo, Palermo, PA
  - AUSL di Piacenza - Ospedale "Guglielmo da Saliceto" di Piacenza, Piacenza, PC
  - Az. ULSS 6 Euganea - Ospedali Riuniti Padova Sud - Ospedale Madre Teresa di Calcutta-Schiavonia, Monselice, PD)
  - Az. ULSS 6 Euganea - Ospedale S. Antonio - Centro Oculistico San Paolo di Padova, Padua, PD
  - A.O. di Perugia - Ospedale S. Maria della Misericordia di Perugia, Perugia, PG
  - Fondazione IRCCS Policlinico S. Matteo - Università degli Studi di Pavia, Pavia, PV
  - Grande Ospedale Metropolitano Bianchi-Melacrino-Morelli di Reggio Calabria, Reggio Calabria, RC
  - Policlinico Universitario Campus Bio-medico di Roma, Roma, RM
  - Fondazione PTV Policlinico Tor Vergata, Roma, RM
  - A.O.U. Sant'Andrea di Roma, Roma, RM
  - IRCCS Fondazione G.B. Bietti di Roma, Roma, RM
  - ASL Roma 4 - Ospedale San Paolo di Civitavecchia, Civitavecchia, RN
  - Az. ULSS 5 Polesana - Ospedale "Santa Maria della Misericordia", Rovigo, RO
  - A.O.U Città della Salute e della Scienza di Torino - Ospedale Molinette, Torino, TO
  - Az. Sanitaria Universitaria Integrata di Trieste - Ospedali Riuniti di Trieste - Ospedale Maggiore, Trieste, TS
  - Az. ULSS 2 Marca Trevigiana - Ospedale di Treviso, Treviso, TV
  - Az. Sanitaria Universitaria Integrata di Udine - P.O. Universitario "Santa Maria della Misericordia" diUdine, Udine, UD
  - Az. ULSS 7 Pedemontana - Ospedale San Bassiano di Bassano del Grappa, Bassano del Grappa, VI
  - Ospedale Sacro Cuore - Don Calabria di Negrar, Negrar, VR
  - A.O.U. Integrata di Verona - Ospedale Borgo Roma, Verona, VR
  - Az. Osp. di Rilievo Nazionale "A. Cardarelli" di Napoli, Napoli
  - A.O.U. "Maggiore della Carità" di Novara, Novara
  - A.O.U. Senese - Università degli Studi di Siena, Siena

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study period:
  * Date of first enrolment: 03.09.2018
  * Date study finalized (LPLV): 19.12.2018
  Study centers:
  * 42 centers in Italy
  * 4 centers in Spain
  * 4 centers in Russia
  * 1 center in Germany
Pre-assignment Details: Planned sample size n.800; randomized patients n.808; screened patients n.863
Groups:
- Levofloxacin + Dexamethasone Followed by Dexamethasone: Levofloxacin + dexamethasone ophthalmic solution containing levofloxacin hemihydrate 5.12 mg/ml, corresponding to levofloxacin 5 mg/ml, and dexamethasone sodium phosphate 1.32 mg/ml, corresponding to dexamethasone 1 mg/ml (L-DSP), followed by Dexamethasone 1 mg/ml ophthalmic suspension (Maxidex)
  Dose and regimen: Levofloxacin + dexamethasone sodium phosphate eye drops for 7 days, 1 x 30 μl drop - 4 times a day, followed by dexamethasone eye drops (Maxidex) for an additional 7 days, 1 drop - 4 times a day.
- Tobramycin + Dexamethasone: Tobramycin 3 mg/ml + dexamethasone 1 mg/ml eye drops suspension (Tobradex)
  Dose and regimen: 1 drop - 4 times a day for 14 days
Period: Overall Study
Arm/Group | Levofloxacin + Dexamethasone Followed by Dexamethasone | Tobramycin + Dexamethasone
Started | 403 | 405
Received at Least One Treatment | 395 | 393
Completed | 388 | 388
Not Completed | 15 | 17
Not completed — Not treated | 8 | 12
Not completed — Treatment and study discontinued | 6 | 2
Not completed — Treatment discontinued + study completed | 1 | 3

BASELINE CHARACTERISTICS:
Population: The analysis population is represented by all randomized patients who received at least one dose of study treatment (Full Analysis Set)
Groups:
- Total: Total of all reporting groups
Arm/Group | Levofloxacin + Dexamethasone Followed by Dexamethasone | Tobramycin + Dexamethasone | Total
Number analyzed (Participants) | 395 | 393 | 788
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 70 | 71 | 141
  >=65 years | 325 | 322 | 647
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.12 (8.55) | 71.84 (8.64) | 71.98 (8.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 229 | 239 | 468
  Male | 166 | 154 | 320
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 0 | 0
  White | 393 | 391 | 784
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Without Signs of Anterior Chamber Inflammation
Description: The number of participants without signs of anterior chamber inflammation (sum of cells and flare score = 0). The following non-inferiority hypotheses has been tested: H0 : πT - πS ≤ - Δ; H1 : πT - πS > - Δ. Where πT and πS are the number of participants without signs of anterior chamber inflammation in the test and standard treatments, respectively, and the non-inferiority margin is Δ = 10%.
Time Frame: Day 15
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Levofloxacin + Dexamethasone Followed by Dexamethasone | Tobramycin + Dexamethasone
Number analyzed (Participants) | 395 | 393
Participants
  Number of participants without signs | 376 | 373
  Number of participants with signs | 19 | 20

2. Secondary Outcome: Number of Participants With Endophthalmitis
Description: The number of participants with endophthalmitis after administration of study treatment in the study was assessed and reported. Diagnosis of endophthalmitis is based on clinical evaluation of signs and symptoms (such as swollen eyelids, ocular pain, conjunctival hyperemia, decreased visual acuity, opaque vitreous) through slit lamp examination, and microbiological tests on conjunctival or corneal swabs.
Time Frame: Day 4, 8, 15
Population: The analysis population is represented by all randomized patients who received at least one dose of study treatment (Full Analysis Set).
  This outcome was not analyzed by applying the Last Observation Carried Forward (LOCF) method to impute missing values if at least one post-baseline value was available.
Measure: Count of Participants; unit: Participants
Arm/Group | Levofloxacin + Dexamethasone Followed by Dexamethasone | Tobramycin + Dexamethasone
Number analyzed (Participants) | 395 | 393
Participants
  Visit 3 - Day 4: no diagnosis of endophthalmitis: number analyzed (Participants) | 393 | 393
  Visit 3 - Day 4: no diagnosis of endophthalmitis | 393 | 393
  Visit 4 - Day 8: no diagnosis of endophthalmitis: number analyzed (Participants) | 391 | 393
  Visit 4 - Day 8: no diagnosis of endophthalmitis | 391 | 393
  Visit 5 - Day 15: no diagnosis of endophthalmitis: number analyzed (Participants) | 389 | 391
  Visit 5 - Day 15: no diagnosis of endophthalmitis | 389 | 391

3. Secondary Outcome: Number of Participants Without Signs of Anterior Ocular Chamber Inflammation
Description: Number of participants without signs of anterior chamber inflammation (sum of cells and flare score = 0).
Time Frame: Day 0 (screening), 4, 8
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Levofloxacin + Dexamethasone Followed by Dexamethasone | Tobramycin + Dexamethasone
Number analyzed (Participants) | 395 | 393
Participants
  Visit 1 - Screening: Number of participants without signs | 395 | 393
  Visit 1 - Screening: Number of participants with signs | 0 | 0
  Visit 3 - Day 4: Number of participants without signs | 289 | 302
  Visit 3 - Day 4: Number of participants with signs | 106 | 91
  Visit 4 - Day 8: Number of participants without signs | 338 | 341
  Visit 4 - Day 8: Number of participants with signs | 57 | 52

4. Secondary Outcome: Conjunctival Hyperemia
Description: Conjunctival hyperemia was evaluated with slit lamp and results provided as a score as follows: 0 = absence of inflammation, 1 = mild inflammation (some vessels injected), 2 = moderate inflammation (diffuse injection of vessels, but individual vessels are still discernable) 3 = severe inflammation (intense injection of vessels, individual vessels not easily discernable).
Time Frame: Day 4, 8, 15
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Levofloxacin + Dexamethasone Followed by Dexamethasone | Tobramycin + Dexamethasone
Number analyzed (Participants) | 395 | 393
Participants
  Visit 3 - Day 4: Score=0 | 337 | 323
  Visit 3 - Day 4: Score>0 | 58 | 70
  Visit 4 - Day 8: Score=0 | 348 | 358
  Visit 4 - Day 8: Score>0 | 47 | 35
  Visit 5 - Day 15: Score=0 | 371 | 375
  Visit 5 - Day 15: Score>0 | 24 | 18

5. Secondary Outcome: Total Ocular Symptoms Score (TOSS)
Description: The TOSS is a patient-reported evaluation in the TOSS Questionnaire of 3 ocular symptoms: itching/burning, hyperemia of conjunctiva and tearing. A score was given in the presence of symptoms: 0 = none, 1 = mild, 2 = moderate, 3 = severe.
Time Frame: Day 4, 8, 15
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Levofloxacin + Dexamethasone Followed by Dexamethasone | Tobramycin + Dexamethasone
Number analyzed (Participants) | 395 | 393
score on a scale
  Visit 3 - Day 4 | 0.29 (0.63) | 0.37 (0.73)
  Visit 4 - Day 8 | 0.28 (0.67) | 0.26 (0.62)
  Visit 5 - Day 15 | 0.17 (0.49) | 0.17 (0.59)

6. Secondary Outcome: Ocular Pain/Discomfort: 4-point Scale
Description: Overall ocular pain and discomfort was evaluated by the subject on a 4-point scale (0 = absent, 1 = mild, 2 = moderate, 3 = severe).
Time Frame: Day 4, 8, 15
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Levofloxacin + Dexamethasone Followed by Dexamethasone | Tobramycin + Dexamethasone
Number analyzed (Participants) | 395 | 393
Participants
  Visit 3 - Day 4: Presence/absence of ocular pain: Score=0 | 360 | 361
  Visit 3 - Day 4: Presence/absence of ocular pain: Score>0 | 35 | 32
  Visit 4 - Day 8: Presence/absence of ocular pain: Score=0 | 366 | 366
  Visit 4 - Day 8: Presence/absence of ocular pain: Score>0 | 29 | 27
  Visit 5 - Day 15: Presence/absence of ocular pain: Score=0 | 377 | 373
  Visit 5 - Day 15: Presence/absence of ocular pain: Score>0 | 18 | 20

7. Secondary Outcome: Use of Rescue Therapy
Description: All rescue therapy used following cataract surgery is to be reported at all visits.
Time Frame: During all the treatment until day 15
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Levofloxacin + Dexamethasone Followed by Dexamethasone | Tobramycin + Dexamethasone
Number analyzed (Participants) | 395 | 393
Participants
  Patients with rescue therapy | 392 | 392
  Patients with no rescue therapy | 3 | 1

8. Other Pre Specified Outcome: Intraocular Pressure (IOP)
Description: IOP is measured using a tonometer. IOP is measured as mmHg; normal intraocular pressures average between 12-22 mm Hg.
Time Frame: At day 0 (screening) and at day 4, 8, 15
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Levofloxacin + Dexamethasone Followed by Dexamethasone | Tobramycin + Dexamethasone
Number analyzed (Participants) | 395 | 393
mmHg
  Visit 1 - Screening | 15.16 (2.48) | 15.12 (2.41)
  Visit 3 - Day 4 | 14.26 (2.73) | 14.49 (2.81)
  Visit 4 - Day 8 | 14.29 (2.51) | 14.45 (3.03)
  Visit 5 - Day 15 | 14.45 (2.65) | 14.37 (2.47)

9. Other Pre Specified Outcome: Visual Acuity
Description: Visual acuity was assessed as per local clinical practice, i.e. with the Snellen (feet) or the ETDRS (meter) chart. Visual acuity was then analysed using decimal unit. Decimal score is the decimal expression of the Snellen (feet) or the ETDRS (meter) charts in which the numerator indicates the distance from the chart and the denominator indicates the size of the smallest line that can be read. Decimal values were provided directly from the investigator or computed as a result of the Snellen or ETDRS fraction.
  Generally decimal values from 0.01 to 0.10 indicate severe vision loss; decimal values from 0.125 to 0.25 indicate moderate vision loss; decimal values from 0.32 to 0.63 indicate mild vision loss; decimal values from 0.8 to 1.6 indicate normal vision.
  Lower decimal values correspond to a reduced visual acuity and worst outcomes, while higher decimal values indicate an improved visual acuity and better outcomes.
Time Frame: At day 0 (screening) and at day 15
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: decimal score
Arm/Group | Levofloxacin + Dexamethasone Followed by Dexamethasone | Tobramycin + Dexamethasone
Number analyzed (Participants) | 395 | 393
decimal score
  Visit 1 - Screening | 0.41 (0.23) | 0.41 (0.26)
  Visit 5 - Day 15 | 0.88 (0.19) | 0.89 (0.17)

10. Other Pre Specified Outcome: Adverse Events
Description: Adverse events were described according to System Organ Classes (SOC) and Preferred Terms (PT) using the Medical Dictionary for Regulatory Activities (MedDRA) and were presented by treatment group.
Time Frame: During all the treatment until day 15
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Levofloxacin + Dexamethasone Followed by Dexamethasone | Tobramycin + Dexamethasone
Number analyzed (Participants) | 395 | 393
Participants
  Patients with TEAEs | 56 | 51
  Patients with serious TEAEs | 4 | 2
  Patients with TEAEs suspected to be study related | 26 | 26
  Patients with TEAEs leading to discontinuation | 4 | 3
  Patients with fatal TEAEs | 1 | 0
  Patients with severe TEAEs | 3 | 0

11. Other Pre Specified Outcome: Global Evaluation of Local Tolerability
Description: Global evaluation was evaluated on a 4-point scale: 0 = no intolerability, 1 = mild intolerability, 2 = moderate intolerability, 3 = maximum intolerability.
Time Frame: Day 4, 8, 15
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Levofloxacin + Dexamethasone Followed by Dexamethasone | Tobramycin + Dexamethasone
Number analyzed (Participants) | 395 | 393
score on a scale
  Visit 3 - Day 4 | 0.03 (0.21) | 0.01 (0.09)
  Visit 4 - Day 8 | 0.01 (0.11) | 0.03 (0.19)
  Visit 5 - Day 15 | 0.02 (0.15) | 0.02 (0.13)

12. Other Pre Specified Outcome: Burning, Stinging, Blurred Vision
Description: Burning, stinging, blurred vision were evaluated on a 4-point scale: 0 = none, 1 = mild, 2 = moderate, 3 = severe.
Time Frame: Day 4, 8, 15
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Levofloxacin + Dexamethasone Followed by Dexamethasone | Tobramycin + Dexamethasone
Number analyzed (Participants) | 395 | 393
score on a scale
  Burning: visit 3 - day 4 | 0.08 (0.27) | 0.09 (0.29)
  Burning: visit 4 - day 8 | 0.06 (0.24) | 0.11 (0.35)
  Burning: visit 5 - day 15 | 0.07 (0.29) | 0.07 (0.27)
  Stinging: visit 3 - day 4 | 0.05 (0.23) | 0.04 (0.20)
  Stinging: visit 4 - day 8 | 0.07 (0.29) | 0.07 (0.26)
  Stinging: visit 5 - day 15 | 0.06 (0.26) | 0.04 (0.20)
  Blurred vision: visit 3 - day 4 | 0.06 (0.27) | 0.05 (0.23)
  Blurred vision: visit 4 - day 8 | 0.06 (0.25) | 0.04 (0.22)
  Blurred vision: visit 5 - day 15 | 0.03 (0.20) | 0.01 (0.11)

13. Other Pre Specified Outcome: Assessment of Patient Diary (Compliance)
Description: Treatment compliance is derived from the number of instillations each day during the study treatment exposure
Time Frame: Day 15
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Levofloxacin + Dexamethasone Followed by Dexamethasone | Tobramycin + Dexamethasone
Number analyzed (Participants) | 395 | 393
Participants
  No missed dose | 332 | 332
  One missed dose per day or three missed doses per | 59 | 57
  > 1 missed dose per day or > 3 missed doses per we | 4 | 4

ADVERSE EVENTS:
Time Frame: From baseline to the end of the treatment, corresponding to 15 days
Description: It is not possible to attribute Adverse Events to Dexamethasone alone following treatment with Levofloxacin + Dexamethasone
Arm/Group | Levofloxacin + Dexamethasone Followed by Dexamethasone | Tobramycin + Dexamethasone
All-Cause Mortality (participants affected / at risk) | 1/395 | 0/393
Serious Adverse Events (participants affected / at risk) | 4/388 | 2/388
Other Adverse Events (participants affected / at risk) | 0/395 | 0/393
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levofloxacin + Dexamethasone Followed by Dexamethasone (N=388) | Tobramycin + Dexamethasone (N=388)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 1 (1)
Retinal Detachment (Eye disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-12): https://cdn.clinicaltrials.gov/large-docs/28/NCT03739528/Prot_SAP_000.pdf